CLINICAL TRIAL: NCT03690479
Title: The Impact of a Modified Probe Tip Design on Patient Perception of Discomfort on Probing and Clinical Parameters Using the Florida Probe® System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Florida Probe Corporation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 244-2011
Record Dates: First submitted 2018-09-25; First posted 2018-10-01 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Periodontitis; Diagnoses Disease
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ball Tip Probe (Active Comparator): One half (upper or lower jaw) of the mouth will be probed using the new trial tip (ball-end probe, 0.6mm diameter).
  Interventions: Device: Ball Tip Probe
- Florida Probe Straight Tip Probe (Active Comparator): One half (upper or lower jaw) of the mouth will be probed using the current, standard probe tip (straight-end probe, 0.45mm diameter).
  Interventions: Device: Florida Probe Straight Tip Probe

INTERVENTIONS:
Device: Florida Probe Straight Tip Probe — Twenty (20) consecutive adult patients with a diagnosis of periodontal disease (varying degrees, from slight to severe) will be selected to undergo full-mouth periodontal probing. . One half (upper or lower jaw) of the mouth will be probed using the current, standard probe tip.
  Other Names: Standard Tip Probe
  Arms: Florida Probe Straight Tip Probe
Device: Ball Tip Probe — Twenty (20) consecutive patients meeting the inclusion criteria will be selected to undergo full-mouth periodontal probing. The opposing jaw will be probed using the new trial tip. At a second visit, prior to treatment, the mouth will be probed once again, alternating the jaws from the first visit.
  Other Names: Titanium Tip Probe
  Arms: Ball Tip Probe

SUMMARY:
Patient perception of pain on periodontal probing using a controlled-force, electronic probe was not significantly affected by the use of a modified (ball-end) probe tip design except for in the maxilla, where a standard straight probe tip appeared to be more comfortable for patients.

DETAILED DESCRIPTION:
Recordings of periodontal probing pocket depth (PPD) and probing attachment level (PAL) are utilized in diagnosis of periodontal disease and monitoring of disease progression. Manual probing presents reproducibility and accuracy issues based on features such as probe tip design, force applied by the operator and inflammatory status of the periodontal tissues. Evidence from the literature suggests that some patients may determine periodontal probing to be a painful experience.

The aims of this study are to evaluate the suitability of a new titanium probe tip for periodontal probing, and to evaluate pain on periodontal probing, in comparison to the existing probe tip used in the Florida Probe® system.

The study will be a randomized, blinded, split-mouth controlled trial. Twenty (20) consecutive patients meeting the inclusion criteria will be selected to undergo full-mouth periodontal probing. One half (upper or lower jaw) of the mouth will be probed using the current, standard probe tip; the opposing jaw will be probed using the new trial tip. At a second visit (within 2 weeks), prior to treatment, the mouth will be probed once again, alternating the jaws from the first visit.

On each occasion, patients will report on pain on probing utilizing two ungraded 100mm horizontal visual analogue scales (VAS) representing upper and lower jaws of the mouth.

Periodontal probing depth measurements will be compared to assess the reproducibility of the two probe tips.

Mean VAS values and standard deviations will be calculated for the test and control groups. Data analysis will be conducted using a non-parametric statistical model (Mann-Whitney U Test).

Inclusion criteria:

* Adult patients: age greater than 18 years.
* At least 4 tooth sites with periodontal probing pocket depth (PPD) greater or equal to 4mm.

Exclusion criteria:

- Patients using ongoing daily chronic analgesic medications (NSAIDs etc) for over 3 months.

ELIGIBILITY:
Inclusion criteria:

* Age greater than 18 years.
* Must have 4 tooth sites with periodontal probing pocket depth (PPD) greater or equal to 4mm.

Exclusion criteria:

- Daily use of analgesic medications (NSAIDs etc) for over 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-04-04 (Actual); Primary Completion 2014-09-06 (Actual); Study Completion 2017-12-14 (Actual)

PRIMARY OUTCOMES:
VAS (visual analogue scale) value 0-100mm | 2 weeks
  Patients will report on pain on probing utilizing two ungraded 100mm horizontal visual analogue scales (VAS): line with values from 0-100, where 0 is no pain and 100 is the worst possible pain, representing upper and lower jaws of the mouth.
  Periodontal probing depth measurements will be compared to assess the reproducibility of the two probe tips.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Harrison, DMD, Principal Investigator — School of Dental Science - Trinity College Dublin
Locations (1):
- University of Florida College of Dentistry, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Canakci V, Canakci CF. Pain levels in patients during periodontal probing and mechanical non-surgical therapy. Clin Oral Investig. 2007 Dec;11(4):377-83. doi: 10.1007/s00784-007-0126-z. Epub 2007 Jun 19. PMID 17576606
- [Background] Fowler C, Garrett S, Crigger M, Egelberg J. Histologic probe position in treated and untreated human periodontal tissues. J Clin Periodontol. 1982 Sep;9(5):373-85. doi: 10.1111/j.1600-051x.1982.tb02048.x. PMID 6754765
- [Background] Hassan MA, Bogle G, Quishenbery M, Stephens D, Riggs M, Egelberg J. Pain experienced by patients during periodontal recall examination using thinner versus thicker probes. J Periodontol. 2005 Jun;76(6):980-4. doi: 10.1902/jop.2005.76.6.980. PMID 15948694
- [Background] Heft MW, Perelmuter SH, Cooper BY, Magnusson I, Clark WB. Relationship between gingival inflammation and painfulness of periodontal probing. J Clin Periodontol. 1991 Mar;18(3):213-5. doi: 10.1111/j.1600-051x.1991.tb01137.x. PMID 2061423
- [Background] Magnusson I, Fuller WW, Heins PJ, Rau CF, Gibbs CH, Marks RG, Clark WB. Correlation between electronic and visual readings of pocket depths with a newly developed constant force probe. J Clin Periodontol. 1988 Mar;15(3):180-4. doi: 10.1111/j.1600-051x.1988.tb01566.x. PMID 3162464
- [Background] Robinson PJ, Vitek RM. The relationship between gingival inflammation and resistance to probe penetration. J Periodontal Res. 1979 May;14(3):239-43. doi: 10.1111/j.1600-0765.1979.tb00229.x. No abstract available. PMID 158084
- [Background] Scott J, Huskisson EC. Graphic representation of pain. Pain. 1976 Jun;2(2):175-84. No abstract available. PMID 1026900
- [Background] Al-Ajmix M, Bogle G, Cole R, Rathbun E, Riggs M, Egelberg J. Ability of examiners to estimate the pain experienced by patients from probing during initial periodontal examination. J Periodontol. 2005 Jun;76(6):985-90. doi: 10.1902/jop.2005.76.6.985. PMID 15948695
- [Background] Chung DT, Bogle G, Bernardini M, Stephens D, Riggs ML, Egelberg JH. Pain experienced by patients during periodontal maintenance. J Periodontol. 2003 Sep;74(9):1293-301. doi: 10.1902/jop.2003.74.9.1293. PMID 14584861